CLINICAL TRIAL: NCT06695884
Title: Determining the Optimal Pulse Protocol for TMS Induced Change in Reward Positivity
Brief Title: Identify the Optimal TMS Pulse Protocol to Modulate Reward Activity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Travis Baker, PhD, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro2022000444_TBSrTMS
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Nicotine Use Disorder
Keywords: transcranial magnetic stimulation; reward processing; EEG; smoking
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single (Participant) Participants will be blinded as to TMS condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Excitatory TMS (Experimental): For condition 1a, 3600 pulses of 10-Hz TMS or 3600 pulses of cTBS. 10 Hz rTMS (110% RMT stimulation intensity; 10 Hz frequency; 5 s on and 26 s off; 3600 pulses per session; total duration of 40 min). cTBS (80% RMT, (3 pulses at 50 Hz with a repeated frequency of 5 Hz, 200 ms intervals, containing 1800 pulses, 60 second break, 1800 pulses; total duration of 5 minutes).
  Interventions: Device: Transcranial Magnetic Stimulation
- Inhibitory TMS (Experimental): For condition 1b, 600 or 1200 pulses of iTBS. iTBS will be administered at 80% of each participant's RMT in a burst-firing pattern (3 pulses at 50 Hz) for a 2 s train, followed by an 8 s period of rest. Across sessions, participants will receive one of two iTBS protocols (randomized): 600 pulses (190 s) or 1200 pulses (570 s).
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — TMS will be delivered using a robotic neuronavigation system (Smartmove, ANT). Stimulation intensity will be standardized. Stimulation will be delivered to the L-DLPFC using a active/placebo figure-8 coil and a magventure TMS device.

SUMMARY:
The primary goal will be to identify the optimal pulse protocol by systematically measuring the efficacy of various theta burst stimulation and repetitive rTMS protocols to increase and decrease the reward positivity in dependent smokers. The secondary objective will be to measure the protocols' effectiveness to increase decision-making capacity using the probabilistic selection task (PST). The third objective will be to specifically assess whether the TMS targets has a differential impact on state levels of craving relative to baseline (Tobacco Craving Questionnaire [TCQ]. The investigators plan to accomplish these three objectives using a randomized, controlled experiment involving 2 sessions.

DETAILED DESCRIPTION:
The design is primarily a randomized control-trial design (2 sessions), comparing the effects excitatory and inhibitory TMS protocols applied to a prefrontal TMS target on reward processing in smokers. Eligible smokers will be invited to attend two experimental sessions over a 1-month period, and asked to abstain from smoking 4 hrs prior to each session. For Sessions A and B, participants will be asked to provide their consent, CO levels and complete the TCQ. Compliance with the 4-hour abstinence period will be defined as breath CO less than 13 ppm. Participants will then be randomly selected to participate in Condition 1a or Condition 1b. All procedures between the two conditions will be identical except for the contrasting TMS protocols (Condition 1a: excitatory protocols, Condition 1b: inhibitory protocols) and the rewards presented in the T-maze task (Condition 1a: monetary rewards, Condition 1b: monetary rewards with cigarette cues). To streamline these studies, the left DLPFC target will be based on conventional DLPFC targeting methods (electrode position F3). For Condition 1a, the protocol administered in Session A and B will be randomized so that participants will either receive 3600 pulses of 10-Hz TMS or 3600 pulses of cTBS. For each session, participants will first engage in one block of T-maze trials (100 trials: Baseline measure). In Condition 1a, participants are told that the reward stimulus indicated 5 cents and that the presentation of the no-reward stimulus indicated the alley was empty (0 cents). Following this block of trials, participants will either receive 10-Hz TMS or cTBS over the predefined DLPFC target (F3), and then asked to complete 3 additional Blocks of the T-maze (300 trials: post-TMS). Immediately after participants complete the T-maze, subjects will be asked to complete the PST and TCQ. At the end of the Session A, participants will complete Session B on a separate day (all procedures identical as Session A). Session A and Session B will be separated by at least 2 days to minimize carryover effects. For Condition 1b, the protocol administered in Session A and B will be randomized so that participants will either receive 600 or 1200 pulses of iTBS. For each session, participants will first engage in one block of T-maze trials (100 trials: Baseline). In Condition 1b, participants are told that the reward stimulus indicated 5 cents and that the presentation of the no-reward stimulus indicated the alley was empty (0 cents). Each reward and no-reward stimulus will be paired with a cigarette cue. Following this block of trials, participants will either receive 600 or 1200 pulses of iTBS over the predefined DLPFC target (electrode F3), and then asked to complete 3 additional Blocks of the T-maze (300 trials: Post-TMS). Immediately after participants complete the T-maze, subjects will be asked to complete the PST and the TCQ. At the end of the Session A, participants will complete Session B on a separate day (all procedures identical as Session A). Session A and Session B will be separated by at least 2 days to minimize carryover effects.

ELIGIBILITY:
Inclusion Criteria:

1. Nicotine dependent individuals (according to the Alcohol, Smoking and Substance Involvement Screening Test nicotine dependence score).
2. Be between the ages of 18 and 55 years old.
3. Not received substance abuse treatment within the previous 30 days.
4. Be in stable mental and physical health.
5. If female, test non-pregnant.
6. No evidence of focal or diffuse brain lesion on MRI.
7. Be willing to provide informed consent.
8. Be able to comply with protocol requirements and likely to complete all study procedures.

Exclusion Criteria:

1. Contraindication to MRI (e.g., presence of metal in the skull, orbits or intracranial cavity, claustrophobia).
2. Contraindication to rTMS (history of neurological disorder or seizure, increased intracranial pressure, brain surgery, or head trauma with loss of consciousness for > 15 minutes, implanted electronic device, metal in the head, or pregnancy).
3. History of autoimmune, endocrine, viral, or vascular disorder affecting the brain.
4. History or MRI evidence of neurological disorder that would lead to local or diffuse brain lesions or significant physical impairment.
5. Life time history of mental disorders such as: Bipolar Affective disorder (BPAD), Schizophrenia, Post-traumatic Stress disorder (PTSD) or Dementia or Major Depression.
6. uninterruptable central nervous system medication

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Event-related Brain Potential: Reward Positivity | Day 0 (day of testing)
  The reward positivity is an event-related brain potential (ERP) sensitive to reward feedback. The reward positivity will be measured during the T-maze task, where participants will receive feedback (Reward, No-reward) following choices. ERPs will be created for each electrode and participant by averaging the single-trial EEG according to feedback type (Reward, No-reward). The reward positivity will be evaluated by subtracting the Reward feedback ERPs from the corresponding No-reward feedback ERPs. The size of the reward positivity will then be determined by identifying the maximum absolute amplitude of the difference wave within a 200-to 400-msec window after feedback onset and evaluated along electrodes Fz, FCz, and Cz. The reward positivity will be measured for each pulse protocol across condition 1a and condition 1b of dependent smokers. The reward positivity will be used to measure the efficacy of the pulse protocol to modulate reward activity.

SECONDARY OUTCOMES:
Approach Learning | Day 0 (day of testing)
  Approach learning will be measured using a Probabilistic Selection task (PST), in which subjects are shown pairs of arbitrary stimuli and must learn by trial-and-error to select one of each pair. During an initial learning phase participants are exposed to three pairs of stimuli, each of the three pairs is rewarded on 80%, 70%, and 60% of the trials. Subjects learn by feedback that some stimuli are associated with more positive feedback (Approach) and that some stimuli are associated with more negative feedback (Avoidance). To determine whether subjects learn more from positive (approach) or negative (avoidance) feedback, during a subsequent testing phase they are required to choose between novel stimulus pairs. Approach learning (accuracy and reaction time) for each proposed pulse protocol across condition 1a and 1b will be measured during the testing phase. Avoidance learning performance will be used to measure the efficacy of the pulse protocol to modulate decision making.

OTHER OUTCOMES:
Nicotine Craving | Day 0 (day of testing - before and after TMS)
  The level of craving will be assessed in dependent smokers using the short version of the Tobacco Craving Questionnaire (TCQ), a 12-item scale that assesses state levels of craving. TCQ will be measured at the start of each session, and following each TMS protocol (once for each pulse protocol). The investigators will compared the TCQ score from pre-TMS (start of session) to post-TMS.

CONTACTS AND LOCATIONS:
Overall Officials: Travis E Baker, PhD, Principal Investigator — Rutgers University
Locations (1):
- Rutgers University - Newark, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Data may be uploaded to an open source framework. All data will be deidentified.